CLINICAL TRIAL: NCT05558501
Title: Intermittent Hypoxia-initiated Plasticity in Humans: A Multi-pronged Therapeutic Approach to Treat Sleep Apnea and Overlapping Co-morbidities
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: John D. Dingell VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PULM-003-22S; CX000125 (Other Grant/Funding Number: eRA)
Record Dates: First submitted 2022-09-19; First posted 2022-09-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Intermittent Hypoxia; Microvascular Function; Fatigability; Maximal Oxygen Consumption; Sympatho-Vagal Balance; CPAP Adherence; Arousal Threshold
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: The present study utilizes a double blind parallel randomized design using an equal allocation ratio for each arm. Block randomization will be conducted to reduce the probability that a disproportionate number of participants are randomized to one group. Mild intermittent hypoxia and "sham MIH" will be administered during wakefulness each day for 15 days over a 3-week period.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study participants will be blinded to the composition of the gas mixture. In addition, the research staff that do not administer the treatment (gas mixture) will complete a blind analysis of all the outcome measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mild Intermittent Hypoxia (MIH) (Experimental): This arm of the protocol will receive mild intermittent hypoxia (8% oxygen) with end-tidal carbon dioxide maintained 2 millimeters of mercury above baseline, while in the laboratory.
  Interventions: Other: Mild Intermittent Hypoxia
- Sham Mild Intermittent Hypoxia (Sham MIH) (Sham Comparator): This arm of the protocol will receive sham MIH (the equivalent of room air), while in the laboratory.
  Interventions: Other: Sham MIH

INTERVENTIONS:
Other: Mild Intermittent Hypoxia — The MIH protocol will be comprised of a 20-minute baseline period followed by exposure to twelve two-minute episodes of hypoxia [partial pressure of end-tidal oxygen (PETO2)= 50 mmHg]. Each episode will be interspersed with a 2-minute recovery period under normoxic conditions. The final episode will be followed by a 30-minute end-recovery period. The partial pressure of end-tidal carbon dioxide (PETCO2) will be sustained 2 mmHg above baseline values for the last ten minutes of baseline and throughout the remainder of the protocol. To rapidly induce a PETO2 of 50 mmHg participants will inspire a gas mixture comprised of 8 % oxygen and 92 % nitrogen from a non-diffusible bag. To maintain PETO2 (i.e. 50 mmHg) and PETCO2 (i.e. 2 mmHg above baseline) at the desired levels supplemental oxygen and carbon dioxide will be added to the inspiratory line from the output of a flow meter device that receives inputs from tanks of 100 % oxygen and 100 % carbon dioxide.
  Arms: Mild Intermittent Hypoxia (MIH)
Other: Sham MIH — During "sham MIH" the participants will be exposed to compressed air (the equivalent of room air).
  Arms: Sham Mild Intermittent Hypoxia (Sham MIH)

SUMMARY:
The prevalence of obstructive sleep apnea (OSA) is high in the United States and is a major health concern. This disorder is linked to numerous heart, blood vessel and nervous system abnormalities, along with increased tiredness while performing exercise likely because of a reduced blood supply to skeletal muscles. The gold standard treatment of OSA with continuous positive airway pressure (CPAP) in many cases does not lead to significant improvements in health outcomes because the recommended number of hours of treatment per night is often not achieved. Thus, development of novel treatments to eliminate apnea and lessen the occurrence of associated health conditions is important. The investigators will address this mandate by determining if repeated exposure to mild intermittent hypoxia (MIH) reduces heart and blood vessel dysfunction and tiredness/ fatigue experienced while exercise performance. The investigators propose that exposure to MIH has a multipart effect. MIH directly targets heart and blood vessel associated conditions, while simultaneously increasing upper airway stability and improving sleep quality. These modifications may serve to directly decrease breathing episodes and may also serve to improve usage of CPAP. Independent of its effect, MIH may serve as an adjunctive therapy which provides another path to reducing heart and blood vessel abnormalities that might ultimately result in improvements in exercise capacity and reverse performance fatigue in individuals with OSA.

DETAILED DESCRIPTION:
The prevalence of obstructive sleep apnea (OSA) is high in the Veteran population and this disorder is linked to numerous cardiovascular, neurocognitive and metabolic abnormalities. Thus, OSA is a major health concern in the Veteran population. Treatment of OSA in many cases does not lead to significant improvements in outcome measures. This inadequacy may be a consequence of reduced treatment adherence with continuous positive airway pressure (CPAP) or because the effect of CPAP on outcome measures is small or absent in some patients despite adequate adherence. Consequently, innovative therapies that directly impact co-morbidities linked to OSA or that increase CPAP adherence could lead to improved outcome measures. In the recent funding cycle, the investigators established that repeated daily exposure to mild intermittent hypoxia (MIH) coupled with CPAP modifies autonomic nervous system activity and dramatically decreases blood pressure compared to CPAP treatment alone. Because MIH was coupled with CPAP, the independent effect of MIH on blood pressure was not established. Moreover, it was not established if these outcomes were sustained for a prolonged time period (i.e. weeks to months).

Although the investigators obtained some indirect evidence that modifications in autonomic nervous system activity were coupled to the reduction in blood pressure, the investigators did not establish if modifications in microvascular function were evident. Microvascular dysfunction together with sympatho-vagal imbalance may have consequences not only for peripheral vascular resistance and blood pressure but also for muscle perfusion and metabolism, thereby limiting exercise performance and increasing fatigability in patients with OSA. Thus, reductions in blood pressure and improvement in microvascular function following treatment with MIH might serve to improve exercise capacity and reverse performance fatigue in individuals with OSA.

Besides its potential effect on autonomic and cardiovascular function, the investigators and others previously established that acute exposure to MIH initiates sustained increases in upper airway muscle activity in humans. This sustained increase is a form of respiratory plasticity known as long-term facilitation. However, in the absence of CPAP the investigators have shown that acute MIH immediately prior to or during sleep leads to increases in apnea severity. This might occur because the manifestation of long-term facilitation is absent in the presence of hypocapnia. Hypocapnia can be induced during sleep by the initiation of another form of plasticity known as progressive augmentation. However, it is possible that the combination of daily exposure to MIH administered many hours before the sleep period may mitigate the effects of progressive augmentation leading to increased upper airway stability.

Independent of this possibility, the investigators showed in the previous funding cycle that increased upper airway stability following treatment with MIH was coupled to a reduction in therapeutic CPAP and improved adherence. However, improved adherence to CPAP might also be linked to an increase in the arousal threshold to both respiratory and non-respiratory stimuli. All the uncertainties outlined above will be addressed in the present proposal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race, 30-60 years of age with a BMI of less than 40 kg/m2 and a weight to hip ratio of less than 1.3in males and 1.2 in females along with pure or predominantly (i.e., comprised of both a central and obstructive component)OSA (AHI less than or equal to 100 events per hour and an average oxygen desaturation level of 85 % or greater).
* Participants will be newly diagnosed and not previously treated with CPAP.
* Participants will also be diagnosed with hypertension. Participants will either be untreated or will be treated unsuccessfully with a single prescribed medication for hypertension. Hypertension will be classified according to the American Heart Association 2018 criteria which includes an elevated systolic blood pressure in the range of 120-129 and a diastolic pressure less than 80 mmHg in addition to stage I and stage II hypertension defined by a systolic blood pressure greater than 130 mmHg and a diastolic pressure greater than 80 mmHg.
* Participants will also be included if they are pre-diabetic (HbA1C: 5.7 - 6.4 %; fasting blood glucose: 100 - 125 mg/dL) and have cholesterol levels ranging from 200-239 mg/dL.
* All participants will have normal lung function and a normal EKG with no or minimal alcohol consumption (< 2 oz of alcohol/night).
* Females will be studied at similar points in their menstrual cycle.

Exclusion Criteria:

* Participants with baseline blood pressure greater than 160/110 will be excluded from participation.
* Participants on any medications, with the exception of a single prescribed medication for individuals with resistant hypertension.
* Participants with any other known disease (e.g. pulmonary hypertension).
* Participants using any sleep promoting supplements including melatonin.
* Night shift workers or participants who recently travelled across time zones.
* Pregnant females.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Pressure | Change at 15 days, 4 and 8- weeks following treatment compared to baseline
  Blood pressure measures over 24 hours will be obtained. Blood pressure will be measured every 20 minutes beginning on Sunday at 6 AM and ending Monday at 6 AM. Participants will wear an actigraph (Actiwatch Spectrum, Respironics) and record their activities in a journal to determine the arousal state (i.e., active wakefulness, quiet wakefulness and sleep) associated with each blood pressure measurement. The data will be separated into active-awake, rest-awake and sleep based on the activity log and corresponding data from an actigraph watch.
  The average value of blood pressure in a healthy individual is 120/80 mmHg. In their participants with OSA, the investigators expect the blood pressure to be higher at baseline and decrease 15 days after treatment. The investigators also expect that this reduction will be maintained at 4 and 8-weeks following treatment.
Change in Microvascular Function (Maximal hyperemic Response) | Change at 15 days, 4 and 8- weeks following treatment compared to baseline
  Microvascular reactivity associated with hyperemia induced by vascular occlusion will be determined by analyzing the maximal hyperemic response (MHR) of tissue saturation index (TSI) signal derived from near-infrared spectroscopy (NIRS) of the lateral gastrocnemius muscle of the non-dominant leg.
  The average value of TSI MHR of the NIRS signals in healthy individuals is 159±9 %. In their participants with OSA, the investigators expect these values to be lower at baseline and to increase 15 days after treatment. The investigators also expect that the increase will be maintained 4 and 8-weeks following treatment.
Change in Microvascular Function (Time to reach Maximal Hyperemic Response) | Change at 15 days, 4 and 8- weeks following treatment compared to baseline
  Microvascular reactivity associated with hyperemia induced by vascular occlusion will be determined by analyzing the time to reach maximal hyperemic response (tM) of tissue saturation index (TSI) signal derived from near-infrared spectroscopy (NIRS) of the lateral gastrocnemius muscle of the non-dominant leg.
  The average value of tM TSI in healthy individuals is 39±5 s. In their participants with OSA, the investigators expect these values to be higher at baseline and to lower 15 days after treatment. The investigators also expect that the decrease will be maintained 4 and 8-weeks following treatment.

SECONDARY OUTCOMES:
Change in Muscle Oxygen Extraction (Time Delay) | Change at 15 days following treatment compared to baseline
  Gastrocnemius muscle deoxygenation will be determined by monitoring temporal variables i.e. time delay of [HHb] signal recorded during the MIH and "sham MIH" treatment. Lying in a supine position, participants will be fitted with the NIRS optode on the belly of the lateral gastrocnemius muscle secured with a double tape or a velcro strap. The NIRS data will be recorded continuously at a sampling rate of 10 Hz and will be analyzed off line.
  The average reported value of [HHb] time delay in a healthy individual is 14.8±1.6s. In their participants with OSA, the investigators expect these values to be higher at baseline and decrease 15 days after treatment.
Change in Muscle Oxygen Extraction (Mean Response Time) | Change at 15 days following treatment compared to baseline
  Gastrocnemius muscle deoxygenation will be determined by monitoring temporal variables i.e. mean response time of [HHb] signal recorded during the MIH and "sham MIH" treatment. Lying in a supine position, participants will be fitted with the NIRS optode on the belly of the lateral gastrocnemius muscle secured with a double tape or a velcro strap. The NIRS data will be recorded continuously at a sampling rate of 10 Hz and will be analyzed off line.
  The average reported value of [HHb] mean response time in a healthy individual is 27.2±2.9s. In their participants with OSA, the investigators expect these values to be higher at baseline and decrease 15 days after treatment.
Change in Sympatho-Vagal Balance (Blood Pressure Variability) | Change at 15 days, 4 and 8- weeks following treatment compared to baseline
  Blood pressure variability will be assessed non-invasively using beat to beat measures of blood pressure. The ratio of low frequency and high frequency range (LF-HF ratio) obtained from the power spectrum analysis of blood pressure variability is considered representative of sympathetic to parasympathetic balance in both physiological and pathophysiological conditions.
  The normal range of LF-HF ratio in a healthy individual is 1.5-2. In their participants with OSA, the investigators expect the ratio to be higher at baseline and decrease 15 days after treatment. The investigators also expect that this reduction will be maintained at 4 and 8-weeks following treatment.
Change in Muscle Oxygen Extraction (Tau) | Change at 15 days following treatment compared to baseline
  Gastrocnemius muscle deoxygenation will be determined by monitoring temporal variable i.e. tau of [HHb] signal recorded during the MIH and "sham MIH" treatment. Lying in a supine position, participants will be fitted with the NIRS optode on the belly of the lateral gastrocnemius muscle secured with a double tape or a velcro strap. The NIRS data will be recorded continuously at a sampling rate of 10 Hz and will be analyzed off line.
  The average reported value of [HHb] tau in a healthy individual is 12.4±2.2s. In their participants with OSA, the investigators expect these values to be higher at baseline and decrease 15 days after treatment.
Change in Maximal Oxygen Consumption | Change at 15 days, 4 and 8- weeks following treatment compared to baseline
  All the participants will complete a maximum oxygen consumption (VO2 max) test using a treadmill. Continuous monitoring of electrical activity of the heart with an electrocardiogram along with the measurement of breath by breath oxygen consumption and carbon dioxide production will be performed.
  The average value of VO2 max in a healthy individual is 35-40 mL/kg/min. In their participants with OSA, the investigators expect the maximal oxygen consumption to be lower at baseline and increase 15 days after treatment. The investigators also expect that this increase will be maintained at 4 and 8-weeks following treatment.
Change in Fatigability | Change at 15 days, 4 and 8- weeks following treatment compared to baseline
  Participants will perform a 10-minute walk test on a 25 m indoor walking course at the beginning and end of the protocol. The distance covered will be recorded every 2.5 minutes and at the end of 10 minutes. The ratio of the average walking speed calculated over the entire 10 minutes of walking and the walking velocity calculated over the first 2.5 minutes of the test will be computed. This ratio will then be normalized to the total distance covered in 10 minutes to calculate the performance fatigability index.
  The average value of performance fatigability index in a healthy individual is less than 1. In the participants with OSA, the investigators expect the performance fatigability index to be higher at baseline and reduce 15 days after treatment. The investigators also expect that this reduction will be maintained at 4 and 8-weeks following treatment.
Change in Sympatho-Vagal Balance (Heart Rate Variability) | Change at 15 days, 4 and 8- weeks following treatment compared to baseline
  Heart rate variability will be assessed non-invasively using beat to beat measures of heart rate. The ratio of low frequency and high frequency range (LF-HF ratio) obtained from the power spectrum analysis of heart rate variability is considered representative of sympathetic to parasympathetic balance in both physiological and pathophysiological conditions.
  The average value of LF-HF ratio in a healthy individual is 1.6±1. In their participants with OSA, the investigators expect the ratio to be higher at baseline and decrease 15 days after treatment. The investigators also expect that this reduction will be maintained at 4 and 8-weeks following treatment.

OTHER OUTCOMES:
Change in CPAP Adherence | Change at 15 days, 4 and 8-weeks following treatment compared to baseline
  CPAP adherence will be assessed by documenting the number of hours of CPAP used per night.
  The average value of CPAP adherence in an individual with OSA is 3.92±0.65 hours per night. In our participants with OSA, the investigators expect the ratio to be lower at baseline and increase 15 days after treatment. The investigators also expect that this increase will be maintained 4 and 8-weeks following treatment.
Change in Arousal Threshold | Change at 15 days, 4 and 8- weeks following treatment compared to baseline
  Arousal threshold to respiratory and non-respiratory (tactile and auditory) stimuli will be measured during baseline polysomnographic and CPAP titration night studies.
  The average value of tone-induced arousal threshold in an individual with OSA is 64.5±2.2 dB. In our participants with OSA, the investigators expect the dB level to be lower at baseline and increase 15 days after treatment. The investigators also expect that this increase will be maintained at 4 and 8-weeks following treatment.
Change in Sleep Apnea Severity | Change at 15 days, 4 and 8-weeks following treatment compared to baseline
  Sleep apnea severity will be determined from the apnea hypopnea index obtained from overnight polysomnographic studies.
  The average value of the apnea hypopnea index in a healthy individual is less than 5 events per hour. In our participants with OSA, we expect the index to be higher at baseline and decrease 15 days after treatment. We also expect that this reduction will be maintained at 4 and 8-weeks following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jason H Mateika, PhD MS BS, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No